CLINICAL TRIAL: NCT03450603
Title: It is Crucial to Identify Predicting Risk Factors for Exacerbation of Chronic Obstructive Pulmonary Disease in Order to Provide Adequate Intensive Therapy and Closer Follow-up
Brief Title: Predicting Risk Factors for Exacerbation of Chronic Obstructive Pulmonary Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-17-019
Record Dates: First submitted 2018-01-23; First posted 2018-03-01 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Investigators will collect the fasting venous blood . White blood cell,C-reactive protein, interleukin-6, -8, -10 and tumor necrosis factor-a will be determined. Sterile swab was used to scratch the oral and buccal mucosa, and gene detection related to chronic obstructive pulmonary disease was conducted to observe whether there were significant differences in the distribution of these genes in different populations.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- stable COPD: Chronic obstructive pulmonary disease (COPD) was confirmed if the patient had a baseline post-bronchodilator FEV1 less than 80% of the reference value and forced expiratory volume in 1 second/forced vital capacity (FEV1/FVC) quotient of less than 70%.Select patients with COPD without acute attack within three months．
- exacerbation of COPD: Exacerbation was defined as an event in the natural course of the disease characterized by a change in the patient's baseline dyspnea, cough, and/or sputum that was beyond normal day to day variations and may have warranted a change in regular medication in a patient with underlying COPD.

SUMMARY:
Exacerbations of chronic obstructive pulmonary disease (COPD) are unfavourable events in the course of disease for most COPD patients. Published evidence indicates a significant impact of exacerbations, especially if frequent, on patients' health-related quality of life (HRQL), disease progression, mortality, health care utilisation and costs. However, the severity,evolution and outcome of an exacerbation may differ significantly between patients - some patients will recover completely in a short period of time while others may die. The identification of risk factors for an adverse outcome could help in distinguishing patients who require more intense management in order to prevent failures, achieve satisfactory recovery and reduce the negative clinical and socioeconomic impact of exacerbations.The pathogenesis of COPD is still unclear, so there is no specific treatment at present .COPD was considered to be the result of a combination of environmental and genetic factors. Genetic factors play an important role in the acute exacerbation of COPD.Therefore, it is an urgent need to explore the heterogeneity of COPD phenotype from the perspective of genes and to seek individualized prevention and treatment programs.This study is intended to provide a theoretical basis for the prevention, evaluation and development of individualized treatment plans for acute exacerbation of COPD, thereby improving the prognosis of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Chronic obstructive pulmonary disease
* aged >= 40 years

Exclusion Criteria:

* spirometry can not be completed because of various reasons
* asthma
* pulmonary embolism
* lung cancer
* sequelae of tuberculosis
* extensive bronchiectasis
* interstitial lung disease
* left cardiac insufficiency

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects aged >40 years,baseline post-bronchodilator FEV1 less than 80% of the reference value and FEV1/FVC of less than or equal to 0.7, when clinically stable or Exacerbation; current,ex-smokers or no smokers. Exclusion Criteria：Participants had COPD complicated by a comorbidity such as pneumothorax, pulmonary embolism, lung cancer, or left cardiac insufficiency. Other exclusion criteria included a diagnosis of asthma, extensive bronchiectasis, sequelae of tuberculosis, interstitial lung disease, or restrictive disease.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-12-10 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with acute exacerbations of chronic obstructive pulmonary disease | one year
  Acute exacerbations of chronic obstructive pulmonary disease is defined as an event in the natural course of the disease characterized by a change in the patient's baseline dyspnea, cough, and/or sputum that is beyond normal day to day variations and may have warranted a change in regular medication in a patient with underlying COPD.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Respiratory Medicine, Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, China